CLINICAL TRIAL: NCT04869189
Title: Non-Invasive Assessment of Contact Lens Performance During Use of a Digital Display
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: CR-6384
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High Sphere (Other): Subjects with a spherical refraction between -1.75 DS and -6.00 DS
  Interventions: Device: JJVC Marketed Contact Lens
- Low Sphere (Other): Subjects with a spherical refraction between -1.50 DS and +1.00 DS
  Interventions: Device: JJVC Marketed Contact Lens

INTERVENTIONS:
Device: JJVC Marketed Contact Lens — Acuvue Oasys® 1-Day
  Other Names: Test 1

SUMMARY:
This is a two-arm, open-label, bilateral dispensing clinical investigation. Eligible subjects will proceed to either a low-sphere or high-sphere arm based on refraction measurements in the baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Between 18 and 35 (inclusive) years of age at the time of screening.
  4. They agree not to participate in other clinical research while enrolled on this study.
  5. They have worn the same brand of soft contact lenses at least eight hours per day for at least two days per week over the previous three months.
  6. They own a wearable pair of spectacles if needed for distance vision correction (by self-report).
  7. They typically use digital devices for a minimum of 4 hours per day, 5 days per week.
  8. In a pre-study screening assessment, they must have a CVS-Q score of 4 or less (asymptomatic group) or 6 or greater (symptomatic group).
  9. They can attain a best-corrected logMAR distance visual acuity of at least 0.20 in each eye.
  10. They have spherical contact lens prescription in the range +1.00 to -6.00 DS (based on the calculated ocular refraction).
  11. They have up to maximum of 0.75 DC of refractive astigmatism (based on the calculated ocular refraction).

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
  3. They have an ocular disorder which would normally contraindicate contact lens wear.
  4. They have had cataract surgery.
  5. They have had corneal refractive surgery.
  6. They are regularly (once per day or more) using oral or inhaled steroids or anti-inflammatory medications.
  7. They are using any topical medications such as eye drops or ointments.
  8. Any known hypersensitivity or allergic reaction to sodium fluorescein.
  9. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear. See section 9.1 for additional details regarding excluded systemic medications.
  10. Participation in any contact lens or lens care product clinical trial within 2 weeks prior to study enrollment.
  11. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  12. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
  13. They have any existing binocular vision anomalies such as strabismus or have been prescribed prisms in their spectacles based on self-report, or in the opinion of the investigator exhibit signs of suppression during binocular vision testing.
  14. Any Efron Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) which in the investigator's opinion would contraindicate contact lens wear.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scales (VAS) | at approximately 2-week follow-up
  Subjective comfort and visual fatigue will be assessed using 0 to 100 on VAS at the start of the visit and at the end of each visual task.
Tear film surface quality | at approximately 2-week follow-up
  Tear film surface quality will be assessed in the left eye (OS) only. The infrared-reflected mires from the tear film will be analyzed using custom image analysis from video recordings. The mean and standard deviation of tear film surface quality metric will be determined across the 5 minutes and at 1-minute increments.
Tear meniscus height | at approximately 2-week follow-up
  The lower tear meniscus in the left eye (OS) only will be analyzed using custom image analysis from video recordings. The mean and SD of tear meniscus height (measured vertically in millimeters) will be determined across the 5 minutes and at 1-minute increments.
Blink frequency | at approximately 2-week follow-up
  Blink frequency will be analyzed using custom image analysis from video recordings. Three blink rate metrics will be determined:
  1. Total blink rate: blinks per minute (all blinks)
  2. Complete blink rate: complete blinks per minute. A complete blink will be defined as having a closed palpebral aperture of less than one third of the open palpebral aperture.
  3. Incomplete blink rate: incomplete blinks per minute. An incomplete blink will be defined as having a closed palpebral aperture of more than one third of the open palpebral aperture.
  Each blink frequency metric will be determined across the 5 minutes and at 1-minute increments.
Interblink interval | at approximately 2-week follow-up
  The distribution of interblink intervals (seconds) over the 5-minute measurement period and at 1-minute increments will be determined in two ways:
  1. Total interblink interval: time in seconds between any blinks
  2. Complete interblink interval: time in seconds between complete blinks
  The number of times the interblink interval exceeds the mean + 1SD tear film break up time (assessed over the extended eye opening periods) will be determined for:
  1. Total interblink interval distribution
  2. Complete interblink interval distribution
Blink completeness | at approximately 2-week follow-up
  The mean and SD of the maximally closed palpebral aperture (in mm) will be summarized for total blinks, complete blinks and incomplete blinks across the 5 minutes. For total blinks, the mean and SD of maximally closed palpebral aperture will also be determined at 1-minute increments.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu